CLINICAL TRIAL: NCT01135212
Title: A Randomized, Double-blind, Candesartan-controlled, Parallel Group Comparison Clinical Study to Evaluate the Antihypertensive Efficacy and Safety of Fimasartan in Patients With Mild to Moderate Essential Hypertension (Phase IIIb)
Brief Title: The Clinical Study to Evaluate the Efficacy and Safety of Fimasartan in Patients With Mild to Moderate Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Kyungpook National University Hospital (Other); Gyeongsang National University Hospital (Other); Keimyung University (Other); Kosin University Gospel Hospital (Other); Daegu Catholic University Medical Center (Other); Dong-A medical center (Unknown); Pusan National University Yangsan Hospital (Other); Yeungnam University Hospital (Other); Ulsan University Hospital (Other); Inje University (Other); Pusan National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A657-BR-CT-302
Record Dates: First submitted 2010-05-31; First posted 2010-06-02 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Hypertension
Keywords: Hypertension; ARB; Fimasartan
MeSH Terms: conditions — Hypertension | interventions — fimasartan; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fimasartan 60mg (Active Comparator): Take one tablet of Fimasartan 60mg once a day in the morning
  Interventions: Drug: Fimasartan 60mg
- Fimasartan 120mg (Active Comparator): Take one tablet of Fimasartan 120mg once a day in the morning
  Interventions: Drug: Fimasartan 120mg
- Candesartan 8mg (Active Comparator): Take one tablet of Candesartan 8mg once a day in the morning
  Interventions: Drug: Candesartan cilexetil

INTERVENTIONS:
Drug: Fimasartan 60mg — Fimasartan 60mg for mild to moderate hypertension. Take a tablet(filled in Doubleblind capsule) every morning.
  Arms: Fimasartan 60mg
Drug: Fimasartan 120mg — Fimasartan 120mg for mild to moderate hypertension. Take a tablet(filled in Doubleblind capsule) every morning.
  Arms: Fimasartan 120mg
Drug: Candesartan cilexetil — Candesartan 8mg for mild to moderate hypertension. Take a tablet(filled in Doubleblind capsule) every morning.
  Other Names: Atacand 8mg
  Arms: Candesartan 8mg

SUMMARY:
The purpose of this clinical study is to evaluate and compare the efficacy and safety of Fimasartan (60mg / 120mg) with Candesartan(8mg) in patients with mild to moderate hypertension.

DETAILED DESCRIPTION:
A randomized, double-blind, Candesartan controlled, parallel group comparison clinical study to evaluate the antihypertensive efficacy and safety of Fimasartan in patients with mild to moderate hypertension Approximately 288 patients will be enrolled in 10 centers in South Korea. This study has planned 5 visits during 14 weeks (placebo run-in period 2 weeks, treatment period 12 weeks). All of the subjects who agreed to participate in this study and gave the written informed consent voluntary are assessed the exclusion and inclusion criteria and receive the investigational product(placebo) at screening visit.

During more than 14 days of placebo run-in period, subjects have to stop the previous anti-hypertension drug. After 2 weeks, subjects are assessed the final eligibility and randomized into one of 3 groups(Fimasartan 60mg, Fimasartan 120mg, Candesartan 8mg) at baseline visit. Subjects take physical and laboratory tests and receive the investigational products per 4weeks during treatment period (12weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who agreed to participate in this study and submitted the written informed consent
2. Subjects aged 19 to 75 years
3. Mild to moderate essential hypertension subjects who are measured more 90mmHg, less than 110mmHg of sitting diastolic blood pressure (SiDBP) at baseline(day 0).
4. Subjects who considered to understand this study , be cooperative, and able to be followed-up whole of the study period.

Exclusion Criteria:

1. Severe hypertension patients; more 110mmHg of SiDBP and/or more 180 mmHg of Sitting systolic blood pressure (SiSBP)
2. Patients with secondary hypertension
3. Patients with significant investigations - abnormal renal function (Creatinine more than upper limit of normal), abnormal liver function (AST, ALT more 2 times than upper normal), moderate fatty lever needed medication
4. Patients with hypotension who has sign and symptom
5. Patients with surgical and medical disease it is able to be affect to absorption, distribution, metabolism, excretion
6. Patients with severe insulin dependent or uncontrolled diabetes mellitus (HbA1c > 9%, regimen change of oral hypoglycemic agent, using insulin)
7. Patients with severe heart disease, ischemic heart disease within 6months, peripheral vascular disease, Percutaneous Transluminal Coronary Angiography (PTCA), Coronary Artery Bypass Graft (CABG)
8. Patients with significant ventricular tachycardia, atrial fibrillation, atrial flutter or other significant arrhythmia
9. Patients with hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, hemodynamically significant aortic valve or mitral valve disease
10. Patients with severe cerebrovascular disease
11. Patients with wasting disease, autoimmune disease, connective tissue disease at present and/or previous.
12. Patients with known severe or malignancy retinopathy
13. Patients with hepatitis B or C or HIV positive reaction
14. Patients who have a story or evidence of alcohol or drug abuse within 2years
15. Patients who are measured the mean difference of mean blood pressure of both arm under SiDBP 10mmHg or SiSBP 20mmHg at screening and baseline visit
16. Patients with history of allergic reaction to any angiotensin II antagonist
17. Patients with any chronic inflammation disease needed to chronic inflammation therapy
18. Childbearing and breast-feeding women
19. Female who plan to become pregnancy or have a possibility of pregnancy but don't prevent conception with acknowledged methods
20. Patients who took medicine within 12 weeks from screening visit or is going on the progress of other clinical trial
21. Subject who are judged unsuitable to participate in this study by investigator

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Sitting Diastolic Blood Pressure | 12weeks from baseline visit
  To compare the difference of Sitting Diastolic Blood Pressure at 12 weeks from baseline visit Fimasartan 60mg with Candesartna 8mg

SECONDARY OUTCOMES:
Sitting DBP | at 12weeks from Baseline visit
  To compare the difference of Sitting Diastolic Blood Pressure at 12 weeks from baseline visit Fimasartan 120mg with Candesartna 8mg
SittingDBP | at 4, 8 weeks from baseline visit
  To compare the difference of Sitting Diastolic Blood Pressure at 4, 8 weeks from baseline visit Fimasartan 60/120mg with Candesartna 8mg
Sitting Systolic Blood Pressure | at 4,8,12 weeks from baseline visit
  To compare the difference of Sitting Systolic Blood Pressure at 4,8,12 weeks from baseline visit Fimasartan 60mg/120mg with Candesartna 8mg
Responder ratio | at 12weeks from baseline visit
  To compare the ratio or responder(SiDBP<90mmHg or difference of SiDBP>10mmHg from baseline) at 12 weeks Fimasartan 60mg/120mg with Candesartna 8mg

CONTACTS AND LOCATIONS:
Overall Officials: ShungChull Chae, Doctor´s degree, Principal Investigator — KuyngPook National Hospital
Locations (1):
- KyungPook National University Hospital, Daegu, Daegu, South Korea

REFERENCES:
- [Derived] Lee JH, Yang DH, Hwang JY, Hur SH, Cha TJ, Kim KS, Kim MH, Chun KJ, Cha GS, Hong GR, Lee SG, Kim DS, Kim DI, Chae SC. A Randomized, Double-blind, Candesartan-controlled, Parallel Group Comparison Clinical Trial to Evaluate the Antihypertensive Efficacy and Safety of Fimasartan in Patients with Mild to Moderate Essential Hypertension. Clin Ther. 2016 Jun;38(6):1485-1497. doi: 10.1016/j.clinthera.2016.04.005. Epub 2016 May 6. PMID 27161546
- [Derived] Fimasartan. Am J Cardiovasc Drugs. 2011 Aug 1;11(4):249-52. doi: 10.2165/11533640-000000000-00000. PMID 21740078